CLINICAL TRIAL: NCT03379935
Title: Radial Head Arthroplasty: A Clinical and Radiological Comparison of Monopolar and Bipolar Radial Head Arthroplasty
Brief Title: Radial Head Arthroplasty A Clinical and Radiological Comparison of Monopolar and Bipolar Radial Head Arthroplasty
Acronym: RHA
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Radial head arthrplasty
Record Dates: First submitted 2017-12-04; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Radial Head Fracture; Elbow Fracture; Arthroplasty Complications
MeSH Terms: conditions — Radial Head and Neck Fractures; Elbow Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bipolar radial head arthroplasty: Patients treated with bipolar head arthroplasty due to radial head fracture
  Interventions: Procedure: Type of radial head arthroplasty
- Unipolar radial head arthroplasty: Patients treated with unipolar head arthroplasty due to radial head fracture
  Interventions: Procedure: Type of radial head arthroplasty

INTERVENTIONS:
Procedure: Type of radial head arthroplasty — Patiens are either treated with a unipolar or a bipolar radial head arthroplasty. At Sundsvall hospital all patients were treated with a unipolar and at Umeå university hospital all patients were treated with a bipolar arthroplasty.

SUMMARY:
Fractures of the radial head are among the most common fractures in the elbow and represent one-third of all elbow fractures.This retrospective cohort study was performed between 2004 and 2014 at Sundsvall and Umeå University hospital, Sweden. All patients who were operated on between 2004 and 2014 with a radial head arthroplasty for an acute or sequelae due to a caput radii fracture.The aim of this study is to evaluate clinical or radiological differences between patients treated with a unipolar or bipolar radial head arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with a radial head arthroplasty during the study period.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with a radial head arthroplasty are included in the study. All patients were asked to participate in the follow-up during 2017.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
QuickDASH | 2-16 years postoperatively
  Patients reported outcome measure. An abbreviated version of the Disabilities the Arm, Shoulder and Hand (DASH) questionnaire. Higher score indicate a greater level of disability, lower scores indicate a lower level of disability. The score ranges from 0 (no disability) to 100 (most severe disability).

SECONDARY OUTCOMES:
Pain | 2-16 years postoperatively
  Visual analogue scale. Range 0-10. Higher value indicate more intensive pain.
Range of motion | 2-16 years postoperatively
  Rang of elbow motion. Measured in grades. Supination, pronation, extension and flexion were measured.
Reoperation | 2-16 years postoperatively
  Number of patients needing revision surgery
Radiographic evaluation | 2-16 years postoperatively
  Radiographic evaluation of the prosthesis. The presence of radiolucent lines, loosening of the prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Bakir Kadum, M.D, Ph.D, Principal Investigator — Umeå University

IPD SHARING:
Plan to Share IPD: Undecided
Researchers are welcome to ask for data. The corresponding author will provide this.

REFERENCES:
- [Background] Heijink A, Kodde IF, Mulder PGH, Veltman ES, Kaas L, van den Bekerom MPJ, Eygendaal D. Radial Head Arthroplasty: A Systematic Review. JBJS Rev. 2016 Oct 18;4(10):e3. doi: 10.2106/JBJS.RVW.15.00095. PMID 27792673
- [Background] Heijink A, Kodde IF, Mulder PGH, Van Dijk CN, Eygendaal D. Cemented bipolar radial head arthroplasty: midterm follow-up results. J Shoulder Elbow Surg. 2016 Nov;25(11):1829-1838. doi: 10.1016/j.jse.2016.05.017. Epub 2016 Aug 9. PMID 27521138
- [Background] Duckworth AD, Wickramasinghe NR, Clement ND, Court-Brown CM, McQueen MM. Radial head replacement for acute complex fractures: what are the rate and risks factors for revision or removal? Clin Orthop Relat Res. 2014 Jul;472(7):2136-43. doi: 10.1007/s11999-014-3516-y. PMID 24549774